CLINICAL TRIAL: NCT04416191
Title: Muscle Immune Cells During Disuse and Recovery in Aging and Metabolic Disease
Brief Title: Immune Cells During Disuse and Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 130232
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Muscle Disuse

STUDY DESIGN:
Intervention Model Description: Participants will be tested before a 2-week limb immobilization period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Limb immobilization (Other): Participants will undergo a 2-week leg immobilization period
  Interventions: Other: Limb immobilization

INTERVENTIONS:
Other: Limb immobilization — Participants will undergo a 2-week period of leg immobilization
  Other Names: Muscle Disuse

SUMMARY:
This is an interventional study enrolling healthy individuals aged 18-35 and 60-85 to understand the recovery of muscle health following a period of inactivity. The enrollment goal is 45 participants. The study will occur over the course of 1-2 months where participants will undergo testing before and after a 2-week limb immobilization period.

DETAILED DESCRIPTION:
Visit 1 (Pre-testing)- After signing a consent form, participants will undergo a blood screening and an oral glucose tolerance test. After the visit, participants will be provided with a step activity monitor to track their level of activity. A dietary assessment will also be determined.

Visit 2- At a later time, the participant will return to the research center for a biopsy, blood draw, body composition scan, MRI and muscle strength testing.

2-week leg immobilization period- After visit 2 , the participant will return home and undergo a 14-day leg immobilization period using the equipment and instructions provided at visit 2.

Visit 3- During the limb immobilization period, participant will return to the research center for a single blood draw.

Visit 4- At the end of the 2-week limb immobilization period, the participant will return to the research center to undergo another biopsy, blood draw, body composition scan, MRI and muscle strength testing.

Visit 5- 2 days after the 2-week limb immobilization period, the participant will return for a biopsy and blood draw.

Visit 6- 7 days after the 2-week limb immobilization period, the participant will be asked to return for a final biopsy, blood draw, body composition scan, MRI and muscle strength testing.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-35 and 60-85 yrs
2. Ability to sign informed consent
3. Free-living, prior to admission

Exclusion Criteria:

* History of cardiovascular disease (e.g., CHF, CAD, right-to-left shunt)
* History of endocrine or metabolic disease such as hypo/hyperthyroidism and diabetes
* History of kidney disease or failure
* Vascular disease
* Risk of DVT including family history of thrombophilia, DVT, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL), and connective tissue diseases (positive lupus anticoagulant), hyperhomocystinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombine III
* Use of anticoagulant therapy (e.g., Coumadin, heparin)
* Elevated systolic pressure >150 or a diastolic blood pressure > 100
* Implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
* Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
* Currently on a weight-loss diet
* Chronic systemic corticosteroid use (≥ 2 weeks) within 4 weeks of enrollment and for study duration (intra-articular/topical/inhaled therapeutic or physiologic doses of corticosteroids are permitted)
* Androgens or growth hormone within 6 months of enrollment and for study duration (topical physiologic androgen replacement is permitted)
* History of stroke with motor disability
* A recent history (<12 months) of GI bleed
* History of liver disease
* History of respiratory disease (acute upper respiratory infection, history of chronic lung disease)
* Pregnancy as determined by a pregnancy test
* Any staff members who report directly to an investigator or who report to someone who reports directly to an investigator.
* Any other condition or event considered exclusionary by the PI and faculty physician

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Thigh Muscle Volume | baseline and after 2 weeks of leg immobilization
  change in thigh muscle volume as determined by MRI
Leg Muscle Strength | baseline and after 2 weeks of leg immobilization
  change in isometric leg extension strength as determined by a isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Micah Drummond, PhD, Principal Investigator — University of Utah
Locations (1):
- The University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
No plan has been put into place